CLINICAL TRIAL: NCT02725164
Title: Anesthetic Gas Leakage in Children During Tonsillectomy: a Comparison of Cuffed and Uncuffed Tracheal Tubes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jerrold Lerman, Clinical Professor of Anesthesia, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Gas leak during tonsillectomy
Record Dates: First submitted 2016-03-25; First posted 2016-03-31 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Exposure to Environmental Pollution; Adverse Effect of Unspecified General Anesthetic
Keywords: oxygen; nitrous oxide; sevoflurane; carbon dioxide; endotracheal tube; respiration
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Uncuffed tracheal tubes (Placebo Comparator): After tracheal intubation with an uncuffed tube, the interventions will be the oxygen concentration, nitrous oxide concentration, carbon dioxide concentration and sevoflurane concentration measured in the tracheal tube compared with those in the oropharynx during spontaneous and controlled ventilation.
  Interventions: Drug: oxygen concentration; Drug: nitrous oxide concentration; Drug: carbon dioxide concentration; Drug: sevoflurane concentration
- Cuffed tracheal tubes (Active Comparator): After tracheal intubation with a cuffed tube, the interventions will be the oxygen concentration, nitrous oxide concentration, carbon dioxide concentration and sevoflurane concentration measured in the tracheal tube compared with those in the oropharynx during spontaneous and controlled ventilation.
  Interventions: Drug: oxygen concentration; Drug: nitrous oxide concentration; Drug: carbon dioxide concentration; Drug: sevoflurane concentration

INTERVENTIONS:
Drug: oxygen concentration — oxygen concentration will be measured in the tracheal tube and oropharynx during spontaneous or controlled ventilation
  Other Names: difference in the oxygen concentration
Drug: nitrous oxide concentration — nitrous oxide concentration will be measured in the tracheal tube and oropharynx during spontaneous or controlled ventilation
  Other Names: difference in the nitrous oxide concentration
Drug: carbon dioxide concentration — carbon dioxide concentration will be measured from the tracheal tube and in the oropharynx during spontaneous or controlled ventilation
  Other Names: difference in the carbon dioxide concentration
Drug: sevoflurane concentration — sevoflurane concentration will be measured in the tracheal tube and oropharynx during spontaneous or controlled ventilation
  Other Names: difference in the sevoflurane concentration

SUMMARY:
Fires and operating room pollution may occur when anesthesia gases leak into the oropharynx during airway surgery. Investigators sought to measure the concentrations of anesthetic gases that leak into the mouth of children undergoing adenotonsillectomy using cuffed and uncuffed tracheal tubes during spontaneous and controlled ventilation.

DETAILED DESCRIPTION:
For the past 6 decades, uncuffed tubes have been used for the children less than 8 years of age out of a fear that cuffed tubes would cause damage to the subglottic region. The correct size uncuffed tube creates a seal in the subglottis that has minimal pressure on the mucosa. However, cuffed tubes have become more widely used in children recently without causing damage to the mucosa. There is very little literature comparing the magnitude of the gas leaks with cuffed and uncuffed tracheal tubes particularly in children. Several authors suggest that the leak of nitrous oxide and sevoflurane with uncuffed tubes was much greater than with cuffed tubes. One important but poorly studied issue is the risk of an airway fire when cautery is used for tonsillectomy because a large leak of oxygen in the mouth could ignite a fire. It also remains unclear whether the mode of ventilation, spontaneous or controlled, affects the leak of gases into the mouth. One might expect that the gas leak with spontaneous ventilation is less than with controlled ventilation, but it may not matter in the context of the small concentrations of oxygen and sevoflurane that investigators use. To address all of these concerns, investigators designed this study to compare the concentrations of gases (oxygen, carbon dioxide, nitrous oxide and sevoflurane) in the oral cavity of children undergoing T&A with either cuffed or uncuffed tubes, during spontaneous and controlled ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. American society of anesthesiologists physical status 1 and 2;
2. fasted
3. scheduled for elective adenotonsillectomy

Exclusion Criteria:

1. refusal of consent by parents
2. difficult tracheal intubation
3. craniofacial anomalies
4. gastroesophageal reflux
5. malignant hyperthermia
6. randomization to a tracheal tube is unacceptable.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Difference in the oxygen concentration with uncuffed and cuffed tubes during spontaneous or controlled ventilation | 8 months
  The differences in the oxygen concentration measured in the trachea and the oropharynx with uncuffed and cuffed tubes during spontaneous or controlled ventilation

SECONDARY OUTCOMES:
Difference in the nitrous oxide concentration with uncuffed and cuffed tubes during spontaneous or controlled ventilation | 8 months
  The differences in the nitrous oxide concentration measured in the trachea and the oropharynx with uncuffed and cuffed tubes during spontaneous or controlled ventilation
Difference in the carbon dioxide concentration with uncuffed and cuffed tubes during spontaneous or controlled ventilation | 8 months
  The differences in the carbon dioxide concentration measured in the trachea and the oropharynx with uncuffed and cuffed tubes during spontaneous or controlled ventilation
Difference in the sevoflurane concentration with uncuffed and cuffed tubes during spontaneous or controlled ventilation | 8 months
  The differences in the sevoflurane concentration measured in the trachea and the oropharynx with uncuffed and cuffed tubes during spontaneous or controlled ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Lerman, MD, FRCPC, Principal Investigator — Women & Children's Hospital of Buffalo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiss M, Dullenkopf A, Gysin C, Dillier CM, Gerber AC. Shortcomings of cuffed paediatric tracheal tubes. Br J Anaesth. 2004 Jan;92(1):78-88. doi: 10.1093/bja/aeh023. PMID 14665558
- [Background] Khine HH, Corddry DH, Kettrick RG, Martin TM, McCloskey JJ, Rose JB, Theroux MC, Zagnoev M. Comparison of cuffed and uncuffed endotracheal tubes in young children during general anesthesia. Anesthesiology. 1997 Mar;86(3):627-31; discussion 27A. doi: 10.1097/00000542-199703000-00015. PMID 9066329
- [Background] Eschertzhuber S, Salgo B, Schmitz A, Roth W, Frotzler A, Keller CH, Gerber AC, Weiss M. Cuffed endotracheal tubes in children reduce sevoflurane and medical gas consumption and related costs. Acta Anaesthesiol Scand. 2010 Aug;54(7):855-8. doi: 10.1111/j.1399-6576.2010.02261.x. Epub 2010 Jun 15. PMID 20560884
- [Background] Mehta SP, Bhananker SM, Posner KL, Domino KB. Operating room fires: a closed claims analysis. Anesthesiology. 2013 May;118(5):1133-9. doi: 10.1097/ALN.0b013e31828afa7b. PMID 23422795
- [Background] Raman V, Tobias JD, Bryant J, Rice J, Jatana K, Merz M, Elmaraghy C, Kang DR. Effect of cuffed and uncuffed endotracheal tubes on the oropharyngeal oxygen and volatile anesthetic agent concentration in children. Int J Pediatr Otorhinolaryngol. 2012 Jun;76(6):842-4. doi: 10.1016/j.ijporl.2012.02.055. Epub 2012 Mar 23. PMID 22444738